CLINICAL TRIAL: NCT05048264
Title: Corticosteroid Injections Administered Under Ultrasound Guidance to Diabetic Patients and the Effect on Blood Glucose
Brief Title: Effect of Corticosteroid Injections on Blood Glucose
Acronym: CSI
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to needed protocol restructuring for study aim expansion and changes to data collection methodology and software model use.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00108093
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus; Steroid Diabetes; Shoulder Osteoarthritis; Knee Osteoarthritis; Adhesive Capsulitis; Hip Osteoarthritis
Keywords: Diabetes; Corticosteroids; Injection; Shoulder; Pain; Osteoarthritis; Knee; Hip
MeSH Terms: conditions — Diabetes Mellitus; Osteoarthritis, Knee; Bursitis; Osteoarthritis, Hip; Pain; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Diabetic patients receiving a corticosteroid injection of their shoulder, knee or hip joints.: There are no study-related interventions for this study.

SUMMARY:
The purpose of this study is to measure the effect of various corticosteroids administered to the shoulder, knee and hip joints in diabetic patients on resultant blood glucose readings.

DETAILED DESCRIPTION:
The purpose of this study is to measure the effect of various corticosteroids administered to the shoulder, knee, and hip joints in diabetic patients on resultant blood glucose readings.

Corticosteroid injections (CSI) are frequently used in orthopedic settings in order to treat a wide array of orthopedic issues, including osteoarthritis, bursitis, tendinitis, and many others. The effect of diabetes on the musculoskeletal system and its role in orthopedic disease has been well-documented. Current evidence demonstrates that corticosteroids, even when administered through a local musculoskeletal injection, can lead to temporary increases in blood glucose. Ultrasound guidance was not explicitly used in any of the studies examining the impact of steroids on blood glucose. The utilization of ultrasound guidance has been shown to increase accuracy when performing injections into the subacromial space as well as the glenohumeral joint when compared to palpation/landmark-guided injections.

ELIGIBILITY:
Inclusion Criteria:

* Known diabetic patients ages 40-75 undergoing clinically indicated standard of care corticosteroid shoulder, knee and hip joint injection
* Ability to perform daily blood glucose testing
* Can receive and send text messages

Exclusion Criteria:

* Previous joint arthroplasty
* Corticosteroid injection at other sites in the body within the past month
* Systemic corticosteroid within the last month other than asthma inhaler
* Anyone who are unable to read and/or understand English
* Pregnant women (self-report)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who has been clinically diagnosed with diabetes and receiving a corticosteroid injection in their shoulder, knee or hip joints.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose measures | Baseline & 2 weeks
  Reported daily glucose measures from baseline to two week after injection

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Ceraulo, MD, Principal Investigator — Duke University
Locations (1):
- Duke Sports Science Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No